CLINICAL TRIAL: NCT01541618
Title: A Longitudinal Study of MSDx Complex 1 as a Marker for Therapy Response in Multiple Sclerosis
Brief Title: A Study of MSDx Complex 1 as a Marker for Therapy Response in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: MSDx, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MSDX-0411
Record Dates: First submitted 2012-02-21; First posted 2012-03-01 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2012-02

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: MS; RRMS; RR Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood remaining after the biomarker test is completed will be retained for possible evaluation of additional biomarkers
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tysabri Group: Patients with a diagnosis of relapsing remitting multiple sclerosis (RRMS) who is about to begin Natalizumab (Tysabri) therapy for a relapse in clinical symptoms (either diagnosed clinically or via gadolinium MRI).
  Interventions: Other: MSDX Complex-1 Biomarker test

INTERVENTIONS:
Other: MSDX Complex-1 Biomarker test — MSDX Complex-1 Biomarker test
  Other Names: Biomarker Test

SUMMARY:
The purpose of this study is to compare biomarker levels in Multiple Sclerosis (MS) patients before and after beginning Natalizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of clinically definite relapsing remitting MS (RRMS)
2. Age 45 years and older
3. Willing and able to provide written informed consent
4. Patient has high disease activity.
5. Patient is about to begin Natalizumab (Tysabri) therapy.

Exclusion Criteria:

1. Any clinically significant disease other than MS that is likely to interfere with the evaluation of CDMS
2. Known infectious or hematological disease.
3. Unwilling or unable to comply with the requirements of this protocol
4. Subject can not have a gadolinium enhanced MRI

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study populations for this study is a patient with a diagnosis of relapsing remitting multiple sclerosis (RRMS) who is about to begin Natalizumab (Tysabri) therapy for a relapse in clinical symptoms (either diagnosed clinically or via gadolinium MRI).
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Change in MSDX Complex-1 between baseline and 6-month visit | 6 months
  This outcome measure will evaluate a difference in the level of MSDX Complex-1 form the baseline visit to the 6-month visit. MSDX Complex-1 is a biomarker for MS disease activity and its change should correspond with a change in the disease activity in MS.

SECONDARY OUTCOMES:
Gadolinium MRI and MSDX Complex-1 level | 6 months
  This outcome will evaluate whether a change seen in a Gadolinium MRI (a diagnostic test for MS) matches with a change in the MSDX Complex-1 level in a patient with MS.

CONTACTS AND LOCATIONS:
Overall Officials: Jeannette Wendt, MD, Principal Investigator — Northwest NeuroSpecialists, PLLC
Locations (1):
- Northwest NeuroSpecialists, PLLC, Tucson, Arizona, United States